CLINICAL TRIAL: NCT00454532
Title: A Phase I/II Clinical Trial Assessing Safety and Efficacy of BZL101 For Metastatic Breast Cancer.
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Bionovo (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: BZL-101-002
Record Dates: First submitted 2007-03-26; First posted 2007-03-30 (Estimated); Results first posted 2012-03-16 (Estimated); Last update posted 2012-03-16 (Estimated); Status verified 2012-02

CONDITIONS: Metastatic Breast Cancer
Keywords: Breast Cancer; Bionovo; BZL101; Chinese Herbs
MeSH Terms: conditions — Breast Neoplasms | interventions — Scutellaria barbata extract

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Drug: BZL101 — Freeze dried powder mixed with liquid. Administered as a daily dose. Dosage to be determined in Phase 1 portion.

SUMMARY:
BZL 101 is an aqueous extract from herba Scutellaria Barbata D. Don of the Lamiaceae family. Preclinical studies suggest that this herb has antitumor activity for breast cancer and preliminary clinical data suggest that it is tolerable in patients with metastatic breast cancer. The overall goals of this Phase I/II trial are to assess the toxicity, maximum tolerated dose, safety and preliminary efficacy of BZL101 for the treatment of advanced metastatic breast cancer.

ELIGIBILITY:
Key Inclusion Criteria:

* Women 18 years or older
* Histologically confirmed breast cancer
* Clinical evidence of metastatic (stage IV) metastasis (other than bone metastasis)
* Availability of estrogen and progesterone receptor status
* At least one measurable disease site defined by RECIST criteria, 30 days prior to study therapy
* For the phase 1, no more that 3 prior cytotoxic regimens for metastatic breast cancer. For the phase 2, no more than 2 prior cytotoxic regimens for metastatic breast cancer
* Life expectancy ≥ 12 weeks
* Eastern Cooperative Oncology Group performance status ≤2
* Women of child bearing potential must agree to 2 forms of contraception during the course of the trial.

Key Exclusion Criteria:

* Inability to understand/unwillingness to sign a written informed consent
* Any significant side effects related to prior chemo, radiation, biology or hormonal therapy that did not resolve in the judgment of the investigator
* Currently using an investigational agent
* Clinically significant gastrointestinal abnormalities
* Currently using coumadin at therapeutic doses or within 2 weeks of taking study medication
* Concurrent palliative radiation or anti-cancer treatment
* Women who report pregnancy, are breast-feeding or have a positive pregnancy test

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 27 (Actual)
Dates: Start 2007-03; Primary Completion 2009-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Deborah Grady, M.D., Principal Investigator — University of California, San Francisco; Charles Shapiro, MD, Principal Investigator — Ohio State University

REFERENCES:
- [Result] Perez AT, Arun B, Tripathy D, Tagliaferri MA, Shaw HS, Kimmick GG, Cohen I, Shtivelman E, Caygill KA, Grady D, Schactman M, Shapiro CL. A phase 1B dose escalation trial of Scutellaria barbata (BZL101) for patients with metastatic breast cancer. Breast Cancer Res Treat. 2010 Feb;120(1):111-8. doi: 10.1007/s10549-009-0678-5. PMID 20054647

RESULTS

PARTICIPANT FLOW:
Groups:
- Level 1: 10g/day
- Level 2: 20g/day
- Level 3: 30g/day
- Level 4: 40g/day
Period: Overall Study
Arm/Group | Level 1 | Level 2 | Level 3 | Level 4
Started | 11 | 6 | 3 | 7
Completed | 11 | 6 | 3 | 7
Not Completed | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Level 1 | Level 2 | Level 3 | Level 4 | Total
Number analyzed (Participants) | 11 | 6 | 3 | 7 | 27
Age Continuous [Median (Full Range); unit: years] | 57 [32 to 78] | 67 [42 to 78] | 55 [54 to 67] | 61 [35 to 66] | 59 [32 to 78]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 11 | 6 | 3 | 7 | 27
  Male | 0 | 0 | 0 | 0 | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2 | 2 | 0 | 1 | 5
  Not Hispanic or Latino | 9 | 4 | 3 | 6 | 22
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0
  Black or African American | 3 | 1 | 1 | 1 | 6
  White | 8 | 5 | 2 | 6 | 21
  More than one race | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 11 | 6 | 3 | 7 | 27

OUTCOME MEASURES:

1. Primary Outcome: Toxicity Based Upon Adverse Events Classifed by the NCI Common Terminology Criteria Version 3 (Phase 1)
Description: Dose-Limiting Toxicities graded according to Common Terminology Criteria for Adverse Events, version 3.0
Time Frame: Monthly
Measure: Number; unit: participants
Arm/Group | Level 1 | Level 2 | Level 3 | Level 4
Number analyzed (Participants) | 11 | 6 | 3 | 7
participants
  Elevated AST | 1 | 0 | 0 | 0
  Diarrhea | 0 | 1 | 0 | 0
  Fatigue | 0 | 1 | 0 | 0
  Pain-rib cage | 0 | 0 | 0 | 1

2. Primary Outcome: Response Evaluation Criteria In Solid Tumors (RECIST) (Phase 2)
Description: Best Overall Tumor Response - Investigator Assessment
Time Frame: 2 Months
Measure: Number; unit: participants
Arm/Group | Level 1 | Level 2 | Level 3 | Level 4
Number analyzed (Participants) | 11 | 6 | 3 | 7
participants
  Complete Response and Partial Response | 0 | 0 | 0 | 0
  Stable Disease | 2 | 3 | 0 | 0
  Progressive Disease | 7 | 3 | 3 | 6
  Unknown | 2 | 0 | 0 | 1

3. Primary Outcome: Response Evaluation Criteria In Solid Tumors (RECIST) (Phase 2)
Description: Best Overall Tumor Response - Independent Radiology Assessment
Time Frame: 2 months
Measure: Number; unit: participants
Arm/Group | Level 1 | Level 2 | Level 3 | Level 4
Number analyzed (Participants) | 11 | 6 | 3 | 7
participants
  Complete Response and Partial Response | 0 | 0 | 0 | 0
  Stable Disease | 3 | 2 | 0 | 1
  Progressive Disease | 0 | 3 | 2 | 3
  Unknown | 8 | 1 | 1 | 3

ADVERSE EVENTS:
Arm/Group | Level 1 | Level 2 | Level 3 | Level 4
Serious Adverse Events (participants affected / at risk) | 5/11 | 0/6 | 1/3 | 4/7
Other Adverse Events (participants affected / at risk) | 11/11 | 6/6 | 3/3 | 7/7
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Level 1 (N=11) | Level 2 (N=6) | Level 3 (N=3) | Level 4 (N=7)
Obstruction-gu ureter (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hemorrhage gu-bladder (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Hemorrhage, GI-abdomen NOS (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pain-breast (Reproductive system and breast disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pain-liver (Hepatobiliary disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hemoglobin (Investigations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Hypoglycemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Thrombosis left iliac vein (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Pain-rib cage due to vomiting (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Infection-ulcer (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Level 1 (N=11) | Level 2 (N=6) | Level 3 (N=3) | Level 4 (N=7)
Nausea (Gastrointestinal disorders) | 4 (4) | 3 (4) | 2 (2) | 5 (5)
Diarrhea (Gastrointestinal disorders) | 5 (6) | 3 (4) | 2 (2) | 5 (5)
Vomiting (Gastrointestinal disorders) | 1 (1) | 2 (3) | 2 (3) | 4 (4)
Fatigue (General disorders) | 1 (1) | 3 (3) | 1 (1) | 3 (3)
Pain-headache (Nervous system disorders) | 3 (3) | 2 (3) | 2 (2) | 1 (1)
Anorexia (Metabolism and nutrition disorders) | 3 (3) | 0 (0) | 0 (0) | 1 (1)
Distension/bloating (Gastrointestinal disorders) | 1 (1) | 2 (2) | 0 (0) | 0 (0)
Flatulence (Gastrointestinal disorders) | 1 (1) | 1 (1) | 0 (0) | 1 (1)
Pain-abdomen NOS (Gastrointestinal disorders) | 2 (2) | 1 (1) | 0 (0) | 1 (1)
Sweating (Skin and subcutaneous tissue disorders) | 2 (2) | 1 (1) | 0 (0) | 1 (1)
Dehydration (Metabolism and nutrition disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
ALT elevation (Investigations) | 3 (3) | 2 (2) | 1 (1) | 0 (0)
AST elevation (Investigations) | 3 (3) | 2 (2) | 0 (0) | 0 (0)
Decreased hemoglobin (Investigations) | 3 (3) | 0 (0) | 1 (1) | 2 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No